CLINICAL TRIAL: NCT04941911
Title: A Double-blind Randomised Placebo-controlled Feasibility Study to Assess the Impact of Octreotide Infusion During Liver Transplantation on Post-operative Renal Failure.
Brief Title: A Feasibility Study of Octreotide Infusion During Liver Transplant.
Acronym: Octreotide
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17/0508; PB-PG-0817-20023 (Other Grant/Funding Number: NIHR Research for Patient Benefit)
Record Dates: First submitted 2021-04-20; First posted 2021-06-28 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Liver Transplantation; Renal Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: Patients will be randomised in a 2:1 ratio to either octreotide or placebo groups. Stratified randomisation of patients by source of liver graft (brain death or cardiac death) will be performed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding (masking) will be achieved through the use of identical active drug product and control study drug syringes that are allocated by centrally-controlled and administered randomisation such that no clinical, research or statistical support staff are aware of allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Octreotide intravenous infusion, 100mcg bolus with a subsequent infusion of 100mcg per hour during surgery.
  Interventions: Drug: Octreotide Acetate
- Placebo group (Placebo Comparator): Sodium chloride 0.9% w/v
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Octreotide Acetate — Octreotide syringes will contain 50ml of octreotide acetate at 20mcg/ml in 0.9% w/v sodium chloride in water.
  Arms: Intervention group
Other: Placebo — Sodium chloride 0.9% w/v
  Arms: Placebo group

SUMMARY:
The purpose of the study is to determine whether an octreotide infusion during liver transplantation improves renal outcomes, intraoperative blood pressure and reduces haemorrhage and transfusion requirement.

DETAILED DESCRIPTION:
Common and serious complications of liver transplantation surgery include renal failure, haemorrhage and blood transfusion. These complications prolong post-operative recovery, increase the risk of liver graft failure, mortality and the need for long-term renal dialysis.

The drug octreotide is a synthetic analogue of somatostatin with comparable physiological effects and a good side-effect profile. Existing evidence in liver transplantation supports octreotide efficacy in improving renal function, reducing bleeding and enhancing blood pressure. However, there is no robust randomised controlled trial evidence for octreotide in liver transplantation and limited safety data regarding its use in this setting.

This is a multi centre, prospective double-blind, randomised, placebo-controlled trial of octreotide infusion during liver transplantation. The patients will be randomised in a 2:1 ratio to either octreotide or placebo groups. Stratified randomisation of patients is by donation type (DCD vs. DBD).

Patients will be randomised in the anaesthetic room and study medication given as an initial bolus of 5ml (100mcg octreotide or saline) prior to surgical incision and then continued throughout surgery at 5ml/hr (100mcg/hour octreotide or saline).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and over undergoing primary liver transplantation of a whole or partial liver graft from a cardiac or brain dead donor.
* Provision of written informed consent.

Exclusion Criteria:

* Previous solid organ transplant.
* Acute liver failure.
* Fulminant hepatic failure.
* Patients receiving a living donor liver graft.
* Patients currently admitted to ICU prior to transplantation.
* Requirement of haemodialysis or CVVHF pre-operatively.
* Known allergy or adverse reaction to octreotide.
* Pre-operative decision to use intra-operative CVVHF.
* A positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Ability to recruit patients. | Approximately 180 days.
  This will be assessed by:
  • Ability to recruit patients (target: ≥ 30% consent rate of eligible patients admitted for transplant)
Completion of the study intervention. | Approximately 9.5 hours.
  This will be assessed by:
  • The percentage of patients successfully completing the study intervention. Defined as eligible patients who receive the entire study drug infusion in a blinded manner.

SECONDARY OUTCOMES:
The incidence of acute kidney injury. | Within 24, 72 and 168 hours post-operatively.
  This will be defined by Acute Kidney Injury Network stage 1 criteria (a 50% increase in serum creatinine from baseline or less than 0.5 ml/kg/hr urine output for 6-12 hours post-transplant).
Post-operative incidence of a new requirement for renal replacement therapy. | Within 24 hours, 72 hours, one and two weeks post-operatively.
  Administration of haemofiltration or haemodiafiltration.
Incidence of new chronic kidney disease or deterioration of chronic kidney disease. | At thirty and ninety days post operative.
  This is defined as a new persistent estimated glomerular filtration rate below 60 ml/min/1.73m2 or a decline in pre-existing glomular function to a more severe KDIGO chronic kidney disease. status.
Incidence of early allograft dysfunction. | At day seven post-operatively
  Early allograft dysfunction defined by the presence of one or more of the following: total bilirubin ≥ 10 mg/dL (171 μmol/L) or, INR ≥ 1.6 on day 7, and ALT/AST > 2,000 IU/L within the first 7 days post-operatively.
Patient mortality. | At thirty and ninety days post-operatively.
  Patient mortality at thirty and ninety days post-operatively.
Intra-operative red blood cell salvage. | Within 24, 72 and 168 hours post-operatively.
  Total volume of intra-operative red blood cell salvage available for reinfusion following washing and centrifugation.
Volume of packed red blood cell transfusion. | Intra-operatively and at 24, 72 and 168 hours post-operatively.
  Volume of packed red blood cell transfusion administered intra-operatively and at 24, 72 and 168 hours post-operatively.
Incidence of adverse events secondary to study drug infusion. | Intra-operatively and up to 24 hours post-operatively.
  Recorded adverse events are: abnormal QTc interval (460ms in men, 470ms in women) or associated ventricular arrhythmia or Torsades de Pointes, unexpected or resistant hypoglycaemia (blood sugar < 4mM) and clinical suspicion of allergic or anaphylactic reaction.
PROMs_ data collection_1 | For EuroQoL-5D-5, At Day 1 and at thirty and ninety days post-operatively. Then at 3, 6 & 9 months.
  PROMs (Patient Recorded Outcome Measures) of quality of life . The questionnaires to be used to quantify quality of life is EuroQoL-5D-5L.
PROMs_ data collection_2 | For LDQOL, At Day 1 and at thirty and ninety days post-operatively. Then at 3, 6 & 9 months.
  PROMs (Patient Recorded Outcome Measures) of quality of life . The questionnaires to be used to quantify quality of life is LDQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Spiro, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - University Hospital Birmingham, Birmingham
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to provide baseline and outcome data, including PROMs and treatment allocation.
Supporting Information: Study Protocol, SAP
Time Frame: Commencement only after publication of this trial and any subsequent substantive trial.
Access Criteria: We would only provide IPD on specific application for that data as part of meta-analysis or other comparable research, rather than providing an 'open book' approach. Eligible requests will come from genuine non-commercial research institutes with a plan to publish meta-analytical or systematic review outcomes. Requests will be reviewed by the TMG with discussion with the TSC as needed. Data will be provided in a basic spreadsheet database via institutional email, ensuring no PID is contained.

REFERENCES:
- [Background] Fabes J, Ambler G, Shah B, Williams NR, Martin D, Davidson BR, Spiro M. Protocol for a prospective double-blind, randomised, placebo-controlled feasibility trial of octreotide infusion during liver transplantation. BMJ Open. 2021 Dec 2;11(12):e055864. doi: 10.1136/bmjopen-2021-055864. PMID 34857585
- [Derived] Coppack KES, Kantsedikas I, Brodkin E, Loh EN, Ambler G, Moonesinghe SR, Fabes J, Hannon V, Spiro M, Wagstaff D. Understanding recruitment to a randomised controlled trial (RCT) during liver transplantation: an observational mixed-methods Study Within A Trial (SWAT). BMJ Open. 2026 Jan 7;16(1):e104310. doi: 10.1136/bmjopen-2025-104310. PMID 41500624